CLINICAL TRIAL: NCT01829815
Title: Impact Evaluation of a Parenting Program to Improve Parenting, Education, and Health Outcomes for Young Children in Liberia
Brief Title: Impact of a Parenting Program in Liberia to Improve Parenting, Education, and Health Outcomes for Children in Liberia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Rescue Committee (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5108
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Parenting Behavior; Pre-academic and Developmental Skills; Malaria Prevention
Keywords: Child; Parents; Parenting; Child Development; Parent Child Relations; Malaria; Primary Prevention; Punishment; Education
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Parents Make the Difference" (Experimental): Caregivers are enrolled in the 10-session Parents Make the Difference intervention.
  Interventions: Behavioral: Parents Make the Difference
- Waitlist Control (Other): Caregivers assigned to the control group received the 10-session Parents Make the Difference intervention after the study was completed.
  Interventions: Behavioral: Parents Make the Difference

INTERVENTIONS:
Behavioral: Parents Make the Difference — The intervention, entitled "Parents Make the Difference," will include 10 sessions. Parents will attend in a group, and sessions will include didactic information, guided discussion, and modeling and practice of new skills. All sessions focus on positive parenting skills, with specific skills across three domains that have strong links to child outcomes: (a) positive, non-physical behavior management strategies, (b) strategies for promoting children's early learning, and (c) strategies, primarily use of bed nets, for preventing malaria in children.

SUMMARY:
The aim of this study is to assess the impact of an intervention to improve parenting practices, pre-academic and developmental skills, and use of mosquito nets for children in kindergarten in Liberia. A rigorous impact evaluation using a randomized, waitlist controlled design will be conducted to measure the impact of the intervention on three primary outcomes: positive parenting skills, children's cognitive and educational skills, and malaria knowledge and prevention behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Parents or primary caregivers (age 18 or above) of children ages 3-7 enrolled in kindergarten
* Resident in one of five study sites

Exclusion Criteria:

* Severe cognitive disability of caregiver affecting ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Parenting Behavior Assessment (adapted from multiple scales for this context) | 1 month
  This is a caregiver-report survey measures including items on various parenting practices, including: caregiver-child communication; discipline and behavior management practices; caregiver-child affection and shared activities; caregiver involvement in child's school and educational activities. These items will yield several subscores for these different domains. Some items may also be analyzed as single items, as they measure specific and important outcomes (e.g., use of a harsh discipline strategy)
Parenting Self-Efficacy and Beliefs Assessment (adapted from other scales for this context; includes unique items developed for this context) | 1 month
  These items assess parents' confidence in their parenting abilities and their beliefs about caregiving practices. This measure will yield separate scores for self-efficacy and beliefs about caregiving practices. Some items may also be analyzed as single items, as they measure specific and important outcomes (e.g., parents' belief about an aspect of harsh discipline)
Child Behavior Assessment (items adapted from the Strengths and Difficulties Questionnaire) | 1 month
  This tool assess children's behaviors and emotional well-being in the domains of hyperactivity, anger, aggression, mood, and peer relationships. They will be analyzed as an overall score, and single items may be analyzed for certain behaviors or indicators of emotional well-being.
Parent-Child Interaction Observation | 1 month
  Caregivers and children in the study will be asked to engage in a play interaction for five minutes, and their verbal interactions will be audio-recorded. Recordings will be coded for specific behaviors. The coding system is adapted from the Dyadic Parent Child Interaction Coding System.
Child Cognitive / Pre-Academic Abilities and Emotional Well-being | 1 month
  Children will be administered activity-based items to assess a range of cognitive and learning skills, including verbal and language skills (as measured by several activities), numeracy, and pattern recognition. Items will be combined into composite scores but may also be analyzed separately to measure outcomes on specific abilities (e.g., counting). Children will also be asked five questions related to their emotional well-being adapted from the Strengths and Difficulties Questionnaire. These items will be analyzed as a sum score, and individual items may be analyzed for specific indicators of emotional well-being.

SECONDARY OUTCOMES:
Mosquito net usage | 1 month
  A survey will be used to assess mosquito net usage by household members. Items will be analyzed separately to assess discrete behaviors (e.g., whether child him/herself slept under the net; whether any adult(s) slept under the net)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Puffer, PhD, Principal Investigator — Duke University; Rhea Chase, PhD, Principal Investigator — Duke University
Locations (1):
- International Rescue Committee, Voinjama, Lofa County, Liberia

IPD SHARING:
Plan to Share IPD: Undecided
File needs to be anonymized

REFERENCES:
- [Derived] Puffer ES, Green EP, Chase RM, Sim AL, Zayzay J, Friis E, Garcia-Rolland E, Boone L. Parents make the difference: a randomized-controlled trial of a parenting intervention in Liberia. Glob Ment Health (Camb). 2015 Aug 4;2:e15. doi: 10.1017/gmh.2015.12. eCollection 2015. PMID 28596863
- [Derived] Annan J, Sim A, Puffer ES, Salhi C, Betancourt TS. Improving Mental Health Outcomes of Burmese Migrant and Displaced Children in Thailand: a Community-Based Randomized Controlled Trial of a Parenting and Family Skills Intervention. Prev Sci. 2017 Oct;18(7):793-803. doi: 10.1007/s11121-016-0728-2. PMID 27858282